CLINICAL TRIAL: NCT01059734
Title: Topoisomerase 2 Expression and Acute Myeloid Leukemia (AML)
Brief Title: S9031-S9126-S9333-S9500-B Biomarker Expression in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S9031-S9126-S9333-S9500-B; S9031-S9126-S9333-S9500-B (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); secondary acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at biomarker expression in bone marrow samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the distributions of topoisomerase 2 (TOP2) expression and single nucleotide polymorphisms (SNPs) in patients with newly diagnosed acute myeloid leukemia (AML).
* Estimate the distributions of mutations in TOP2 phosphorylation sites (by SNP analysis) in these patients.
* Investigate whether expression of TOP2 or mutations in TOP2 phosphorylation sites vary with patient or disease characteristics in these patients.
* Test whether TOP2 expression correlates with complete remission rates, relapse-free survival, and overall survival of these patients.
* Conduct preliminary analyses to estimate the distributions of TOP2 expression and mutations in TOP2 phosphorylation sites (by SNP analysis) in patients with relapsed and/or refractory AML.
* Investigate whether expression of TOP2 and mutations in TOP2 phosphorylation sites vary with patient or disease characteristics in patients with relapsed and/or refractory AML.
* Test whether TOP2 expression and mutations in TOP2 phosphorylation sites differ between previously untreated and relapsed/refractory AML patients.

OUTLINE: This is a multicenter study.

Archived RNA specimens are analyzed for topoisomerase 2 transcriptional expression by quantitative real-time polymerase chain reaction (PCR) and for mutations within TOP2 phosphorylation sites by single nucleotide polymorphism analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia

  * All subtypes allowed (except acute promyelocytic leukemia [M3])
  * Previously untreated OR relapsed/refractory disease
* Isolated RNA specimens from bone marrow aspirate samples available from patients who participated on SWOG-9031, SWOG-9333 (cytarabine/daunorubicin hydrochloride induction arm only), SWOG-9500, or SWOG-9126

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enrolled on S0931, S9126, S9333 or S9500 consenting to use of specimens for future research
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Distribution of topoisomerase 2 (TOP2) expression and single nucleotide polymorphisms | immediate
Distributions of mutations in TOP2 phosphorylation sites | immediate
Correlation of TOP2 expression with complete remission rates, relapse-free survival, and overall survival | immediate
Variation of TOP2 expression and mutations in TOP2 phosphorylation sites among patients and disease characteristics | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Principal Investigator — The Cleveland Clinic

REFERENCES:
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844